CLINICAL TRIAL: NCT00075894
Title: A Phase I/II, Open-Label, Non-Randomized, Multicenter, Single Agent Study Of Intravenous SDX-102 For The Treatment Of Patients With MTAP-Deficient High Grade Recurrent Malignant Gliomas
Brief Title: Alanosine in Treating Patients With Progressive or Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000349473; NABTT-0303
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2006-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic oligodendroglioma; adult anaplastic astrocytoma; adult glioblastoma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Astrocytoma; Glioblastoma; Brain Neoplasms; Gliosarcoma | interventions — alanosine

INTERVENTIONS:
Drug: L-alanosine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as alanosine, use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of alanosine in treating patients with high-grade progressive or recurrent malignant gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of alanosine (SDX-102) with or without enzyme-inducible antiepileptic drugs (EIAEDs) in patients with methylthioadenosine phosphorylase (MTAP)-deficient high-grade progressive or recurrent malignant gliomas.
* Determine the pharmacokinetics of this drug administered concurrently with EIAEDs in these patients.

OUTLINE: This is an open-label, nonrandomized, multicenter, dose-escalation study. Patients are stratified according to concurrent anticonvulsant drug use (drugs that induce hepatic metabolic enzymes vs drugs that cause modest or no induction of hepatic metabolic enzymes OR no anticonvulsant drug).

Patients receive alanosine (SDX-102) IV continuously for 5 days. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SDX-102 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study therapy, patients are followed at 1 week and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant glioma of 1 of the following types:

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Progressive or recurrent disease after prior radiotherapy with or without chemotherapy

  * Low-grade glioma that progressed after prior radiotherapy with or without chemotherapy and is found to be high-grade glioma after biopsy allowed
  * No more than 2 prior treatment regimens
* Measurable disease by CT scan or MRI
* Documented absence of methylthioadenosine phosphorylase (MTAP) on fixed tumor specimens

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* Transaminases ≤ 4 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception before, during, and for 4 weeks after study participation
* Mini mental state exam score of ≥ 15
* No psychological or sociological condition, addictive disorder, or family problem that would preclude study compliance
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* No concurrent serious infection or medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy

* Must be maintained on a stable or lower corticosteroid regimen from the time of the baseline scan until the start of study treatment
* No concurrent steroids as antiemetics

Radiotherapy

* See Disease Characteristics
* At least 3 months since prior radiotherapy

Surgery

* Not specified

Other

* Recovered from prior therapy
* More than 10 days since prior anticonvulsant drugs that induce hepatic metabolic enzymes
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Surasak Phuphanich, MD, FAAN, Study Chair — Emory University
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina